CLINICAL TRIAL: NCT04558190
Title: Mitochondrial Dysfunction and Insulin Resistance in Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: mtROS-IR
Record Dates: First submitted 2020-09-02; First posted 2020-09-22 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — soybean oil, phospholipid emulsion; mitoquinone; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lipid infusion + MitoQ (Experimental): Subjects undergo a hyperinsulinemic isoglycemic clamp preceded by MitoQ administration and intravenous lipid infusion
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion; Dietary Supplement: MitoQ
- Lipid infusion + placebo (Placebo Comparator): Subjects undergo a hyperinsulinemic isoglycemic clamp preceded by placebo administration and intravenous lipid infusion
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion
- Control (No Intervention): Subjects undergo a hyperinsulinemic isoglycemic clamp
- Lipid infusion + beta2-agonist (Other): Subjects undergo a hyperinsulinemic isoglycemic clamp with intravenous infusion of lipid and salbutamol
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion; Drug: Salbutamol

INTERVENTIONS:
Drug: Intralipid, 20% Intravenous Emulsion — Lipid infusion
  Arms: Lipid infusion + MitoQ; Lipid infusion + beta2-agonist; Lipid infusion + placebo
Dietary Supplement: MitoQ — Oral administration of MitoQ capsules
  Other Names: Mitoquinone mesylate; Mitoquinone; MitoQ10
  Arms: Lipid infusion + MitoQ
Drug: Salbutamol — Beta2-agonist infusion
  Arms: Lipid infusion + beta2-agonist

SUMMARY:
The purpose of the study is to evaluate the link between insulin resistance and alterations in skeletal muscle mitochondrial redox homeostasis

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥25 and <40 kg/m2
* Fasting plasma glucose ≥ 5.6 mmol/L or HbA1c ≥ 5.7%
* HOMA2-IR > 1.4
* VO2max <45 ml/kg/min

Exclusion Criteria:

* Treatment with >2 antidiabetic medications
* Insulin usage
* Chronic disease deemed by the study responsible medical doctor to interfere with any part of the study
* Chronic use of prescription medicine deemed by the study responsible medical doctor to interfere with any part of the study
* Smoking

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Whole body Insulin sensitivity | 5 hours after lipid infusion
  Whole body insulin sensitivity is determined by hyperinsulinemic isoglycemic clamp method
Skeletal muscle insulin sensitivity | 5 hours after lipid infusion
  Insulin-dependent skeletal muscle glucose uptake is determined by hyperinsulinemic isoglycemic clamp method integrated with measurements of femoral artery blood flow and arteriovenous difference of glucose

SECONDARY OUTCOMES:
Mitochondrial respiration | Baseline
  Mitochondrial O2 flux is determined in skeletal muscle biopsies by high-resolution fluorespirometry
Mitochondrial reactive oxygen species | Baseline
  Mitochondrial H2O2 emission rate is determined in skeletal muscle biopsies by high-resolution fluorespirometry
Mitochondrial oxidative stress | Before (baseline) as well as 3 and 5 hours after lipid infusion
  Peroxiredoxin3 dimer/monomer ratio is determined in skeletal muscle biopsies
Muscle redox status | Before (baseline) as well as 3 and 5 hours after lipid infusion
  GSH/GSSG ratio is determined in skeletal muscle biopsies
Insulin signalling | Before (baseline) as well as 3 and 5 hours after lipid infusion
  Phosphorylation status of proteins modulating insulin action is determined in skeletal muscle biopsies

OTHER OUTCOMES:
Cardiorespiratory fitness | Baseline
  Pulmonary maximal oxygen uptake (VO2max) is determined during an incremental exercise test to exhaustion
Body composition | Baseline
  Fat free mass and fat mass are determined by dual-energy X-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No